CLINICAL TRIAL: NCT05473468
Title: A Single Center, Single Dose, Open Label Phase 1 Study To Evaluate The Pharmacokinetics, Excretion, Mass Balance And Metabolism Of [14c]-Famitinib In Healthy Adult Male Subjects
Brief Title: Single Dose Study To Study The Absorption, Metabolism And Excretion Of Famitinib
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-107
Record Dates: First submitted 2022-07-20; First posted 2022-07-26 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — famitinib

STUDY DESIGN:
Intervention Model Description: Single oral dose of [14c]-Famitinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: Famitinib

INTERVENTIONS:
Drug: Famitinib — a single oral dose of [14C]famitinib (25 mg/150 uCi suspension)

SUMMARY:
The purpose of this study is to evaluate the excretion balance, metabolic profile and the routes of excretion of famitinib in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male between the ages of 18 and 45 years;
2. Total body weight ≥ 50 kg, and the Body Mass Index (BMI) of 19 to 28 kg/m2;
3. Male subjects of childbearing potential and their partners have no birth or sperm donation plan and voluntarily take effective contraception during the course of clinical trial until 6 months after the drug administration;
4. An informed consent document signed and dated by the subject;
5. Normal bowel movements (1 to 2 times a day), no habitual constipation or diarrhea.

Exclusion Criteria:

1. No clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests;
2. Positive results of hepatitis B surface antigen, hepatitis C antibody, HIV antibody or treponema pallidum antibody;
3. Have taken any clinical trial drug or participated in any clinical trial within 3 months before administration;
4. CYP3A4 inducers or inhibitors were taken within 28 days before administration;
5. Have taken any prescription or over-the-counter drugs, vitamin products, health care drugs, traditional Chinese medicines or food supplements within 14 days before administration;
6. Those who need to receive anticoagulant therapy such as warfarin or thrombin inhibitors and/or aspirin antiplatelet therapy within 1 month before administration and during the study period;
7. There are clinically significant bleeding symptoms or clear bleeding tendencies within 3 months before administration, such as gastrointestinal bleeding and peptic ulcers;
8. History of stroke or intracranial hemorrhage within 6 months before administration;
9. Have uncontrolled clinical symptoms or diseases of the heart, such as: (1) heart failure above NYHA2 (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) screening period QTcF >450 ms (male);
10. Those who have undergone major surgery within 6 months before administration or that surgical incision has not completely healed; Major surgery includes, but is not limited to, any surgery that is at significant risk of bleeding, prolongs the period of general anesthesia, or has an incision biopsy or significant traumatic injury;
11. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before administration;
12. Hemorrhoids or perianal diseases accompanied by regular / hematochezia; Those with gastrointestinal abnormalities such as irritable bowel syndrome and inflammatory bowel disease, which may affect drug absorption as determined by investigator;
13. People with allergic constitution or allergic diseases, including those with severe drug allergies or history of drug allergies, and those who are known to be allergic to famitinib or excipients;
14. Have any history of clinical serious diseases or diseases or conditions that the researcher believes may affect the results of the trial, including but not limited to circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, psychiatric and metabolic disease history; Lifestyle Habits;
15. History of alcoholism with alcohol consumption over 14 units per week;; and can't abstain from smoking and alcohol during the study;
16. Heavy smoker or habitually use nicotine-containing products;
17. Have a history of drug abuse or have used soft drugs (such as: marijuana) within 3 months before administration or take drugs (such as cocaine, amphetamines, phencyclidine, etc.) within 1 year before administration; or positive urine drug abuse test during screening periods;
18. Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages (more than 8 cups a day, 1 cup = 250 mL) and unable to quit during the study period;
19. Those who cannot tolerate venipuncture or with a history of needle-sickness and blood-sickness;
20. Workers who require long-term exposure to radioactive conditions; or those who have significant radiation exposure (≥ 2 chest/abdominal CT scans, or 3 other X-ray tests ≥) within 1 year prior to administration or who have participated in radiopharmaceutical labeling tests;
21. Blood donation no less than 400 mL or have blood transfusion within 3 months of dosing;
22. Subjects who, in the opinion of the Investigator should not participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta urine: CumAe and Cum%Ae | 0-336 hours
  Amount and cumulative amount excreted and expressed as the percentage of the administered dose into the urine from time t1 to time t2
Mass balance recovery of total radioactivity in all excreta feces: CumAe and Cum%Ae | 0-336 hours
  Amount and cumulative amount excreted and expressed as the percentage of the administered dose into the feces from time t1 to time t2
Total recovery of radioactivity in urine and feces as percentage of total radioactive dose administered | 0-336 hours
  To characterize the extent of excretion of total radioactivity in urine and feces following administration of famitinib
Metabolic Profiling in Blood | 0 to 240 hours
  Metabolic profiling/identification and determination of relative abundance of famitinib and the metabolites of famitinib in plasma if possible.
Metabolic Profiling in Urine | 0-336 hours
  Metabolic profiling/identification and determination of relative abundance of famitinib and the metabolites of famitinib in urine if possible.
Metabolic Profiling in Feces | 0-336 hours
  Metabolic profiling/identification and determination of relative abundance of famitinib and the metabolites of famitinib in feces if possible.
Ratio of radioactivity of whole blood and plasma blood | 0-72 hours
Radioactivity AUC | 0-240 hours
Plasma famitinib and SHR116637: AUC | 0-240 hours
Plasma famitinib and SHR116637: Cmax | 0-240 hours
Plasma famitinib and SHR116637: Tmax | 0-240 hours
Radioactivity Tmax | 0-240 hours
Radioactivity Cmax | 0-240 hours
Plasma famitinib and SHR116637: t1/2 | 0-240 hours
Radioactivity t1/2 | 0-240 hours

SECONDARY OUTCOMES:
AEs and SAEs | 0-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided